CLINICAL TRIAL: NCT04885803
Title: Vitamin D Absorbance Study - A Decentralized, Randomized, Double-blind, Placebo-controlled Clinical Trial of the Pharmacokinetics of Vitamin D3 Absorption From Softgel Supplements Compared to Nano Liquid D3 Supplements in Humans.
Brief Title: Vitamin D Absorbance Study - Clinical Trial of the Absorbance of Nano Liquid D3
Acronym: ViDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inspired Life Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Vitamin D Absorbance Study
Record Dates: First submitted 2021-05-06; First posted 2021-05-13 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Full blinding protocols employed to mask all participants, all those engaging with participants, and the PI for the duration of the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nano Liquid D3 (Experimental): Arm receiving Nano Liquid Vitamin D3
  Interventions: Dietary Supplement: Nano Liquid Vitamin D3; Diagnostic Test: 25(OH)D Blood Serum Test
- Softgel D3 (Active Comparator): Group receiving Softgel Vitamin D3
  Interventions: Dietary Supplement: Softgel Vitamin D3; Diagnostic Test: 25(OH)D Blood Serum Test
- Placebo Control (Placebo Comparator): Liquid mixture, identical in process, taste, smell, and appearance to Nano Liquid D3, but containing no active ingredient (no Vitamin D3)
  Interventions: Diagnostic Test: 25(OH)D Blood Serum Test; Other: Placebo Control

INTERVENTIONS:
Dietary Supplement: Softgel Vitamin D3 — 5000IU vitamin D3 taken as single oral softgel once daily for 30 days
  Other Names: Cholecalciferol
  Arms: Softgel D3
Dietary Supplement: Nano Liquid Vitamin D3 — 5000IU vitamin D3 taken as liquid oral spray once daily for 30 days
  Other Names: Cholecalciferol
  Arms: Nano Liquid D3
Diagnostic Test: 25(OH)D Blood Serum Test — A sample of blood is drawn off and processed for 25(OH)D levels at baseline, after 15 days of supplementation, and after 30 days of supplementation
  Other Names: Vitamin D Blood Test
Other: Placebo Control — Liquid oral spray once daily for 30 days. Solution identical in smell, taste, color, and production process to Nano Liquid D3, but containing no Vitamin D3.
  Other Names: Nano Liquid Placebo
  Arms: Placebo Control

SUMMARY:
Vitamin D is a commonly available essential prohormone humans need to regulate blood calcium and has recently emerged as potentially helpful in combating severe COVID-19. Despite its importance, some studies estimate as much as 40% of the US population is deficient in vitamin D. Most available vitamin D supplements have little absorption data and are nearly all softgels or capsules. This clinical trial is designed as a preliminary pharmacokinetics study to assess the absorbance of a nano liquid D3 supplement that can be taken as an oral spray once daily. Preliminary evidence suggests that this nano liquid D3 may be absorbed more readily than commercially available softgel dosage forms of D3. This randomized, double-blind, placebo-controlled trial will compare nano liquid D3 to commonly available D3 oral softgels and a placebo control group over the course of a thirty-one (31) day study period.

ELIGIBILITY:
Inclusion Criteria:

* Adults, ages 18-70 years old
* Either male or female
* Taking less than 2,000 IU of vitamin D daily as a supplement during the 30 days before starting the study
* Ability to swallow a pill of typical size or a liquid less than 1 mL daily for 30 days
* Ability to speak, read, and understand English
* Access to smart phone or smart device with internet access for study-related communications
* Ability to do 3 at-home vitamin D finger prick blood tests on 3 separate days. The kits and supplies will be given to you.
* Ability to drop off finished blood tests at a UPS store or UPS drop box, or schedule a UPS pickup at your home, on each of the same days as you do the blood tests

Exclusion Criteria:

* Females who are pregnant
* Taking, on average, more than 2,000 IU of vitamin D daily within 30 days before the study
* Currently have COVID-19 infection
* History of COVID-19 infection or positive COVID-19 test in last 60 days
* People with a diagnosis of Cystic Fibrosis
* People with a diagnosis of Crohn's Disease
* People diagnosed with Celiac Disease
* People with known diagnosis or history of any kidney related disease Including, but not limited to: Chronic kidney disease; End stage renal disease; Polycystic kidney disease; Lupus nephritis; Kidney cancer, Alport syndrome; Amyloidosis; Goodpasture syndrome; and Wegener's granulomatosis
* People with known diagnosis or history of any liver related disease Including, but not limited to: Hepatitis A; Hepatitis B; Hepatitis C; Fatty liver disease; Cirrhosis of the liver; Liver cancer; Hemochromatosis; Wilson disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in 25(OH)D Blood Serum Levels | 31 days
  Change in 25(OH)D blood serum levels in the test group taking 5,000 IU of Nano Liquid D3 daily after supplementation compared to the placebo control during the same time frame

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Schroeder, PharmD, Principal Investigator — Inspired Life Medical, Inc.; Noah B Goodson, PhD, Study Director — The Scope Method, LLC
Locations (1):
- Inspired Life Medical Office, Le Sueur, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided